CLINICAL TRIAL: NCT05058430
Title: SaliPen Human Factors Study for OTC Labeling
Acronym: SaliPen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saliwell Ltd. (Industry)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IU12473
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-06

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subjects with xerostomia (Experimental): The primary objective of this research is to assess the human factors in relabeling the SaliPen from a prescription-based device to an OTC.
  Primary performance endpoints:
  * The user can select the device properly.
  * The user can use the device as instructed in the IFU.
  Interventions: Device: Electrical salivary stimulator system assigned to subjects with xerostomia
- Subjects without xerostomia (Active Comparator): The primary objective of this research is to assess the human factors in relabeling the SaliPen from a prescription-based device to an OTC.
  Primary performance endpoints:
  • The user can select the device properly.
  Interventions: Device: No Electrical salivary stimulator system assigned to subjects without xerostomia

INTERVENTIONS:
Device: Electrical salivary stimulator system assigned to subjects with xerostomia — SaliPen is an electrical salivary stimulator system, intended to electrically stimulate a relative increase in saliva production. It is an intraoral device indicated for use in patients with xerostomia (dry mouth).
  Arms: Subjects with xerostomia
Device: No Electrical salivary stimulator system assigned to subjects without xerostomia — SaliPen is an electrical salivary stimulator system, intended to electrically stimulate a relative increase in saliva production. It is an intraoral device indicated for use in patients with xerostomia (dry mouth).
  Arms: Subjects without xerostomia

SUMMARY:
This Human Factors Validation Testing will assess user interactions to verify the capability of potential users to assess if the study product fits their needs and if they can use it correctly based on the provided Information For User (IFU)?

More specifically, this is a non-comparative case series study and is subdivided into two major parts. Those parts are:

1. Phase I: aimed at testing if, based on the IFU, the potential subjects can decide whether the study product is or is not appropriate to treat their condition and,
2. Phase II: aimed at assessing whether the users can use the study product correctly without counseling by a health care provider.

DETAILED DESCRIPTION:
Phase I To simulate an OTC setting, potential subjects will be requested to read the label text on the outside of the study product package (external labeling) and determine whether the study product addresses their needs, without a provider direction or assistance.

Phase II The study product will be dispensed only to those subjects who will indicate that they voluntarize to participate in this phase of the study.

At Phase II subjects with xerostomia and that are willing to try the study product, will be requested to use it with no training, except for their understanding of the User Manual (internal labeling). Those subjects will use the study product in a supervised clinical setting. Subjects who report any discomfort will be offered the option to pause and remove the device upon such a request.

Correct use verification will be performed by the study investigators. Subjects will answer questions regarding product use, clarity of the IFU, ease of use, etc. Subjects will also receive an exam of their oral cavity.

ELIGIBILITY:
Inclusion Criteria:

For Phase I: 8 subjects with xerostomia and 8 without that are 18 years old or older For Phase II: Subjects with xerostomia that are 18 years old or older

Exclusion Criteria:

For Phase I:

* Children and adolescents (persons under 18 years of age)
* Persons with experience in the use of SaliPen

For Phase II: Subjects for them the study product is not indicated and/or do not agree to participate in Phase II. For the avoidance of doubt, the following conditions are exclusion criteria:

* Persons with experience in the use of SaliPen
* Children and adolescents (persons under 18 years of age)
* Epileptic disorder
* Persons that are allergic to the surface materials of the device

  * Electrodes: coated with gold
  * Body: made of methyl vinyl silicone rubber
* Use of a pacemaker
* Pregnancy
* Psychiatric or psychological disorders
* Involuntary muscle movement disorder (such as Parkinson's)
* Neurologic disorder in head and neck area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Zunt, DDS, MS, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Dentistry, Oral Health Research Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients visiting the participating clinic were asked to participate in the study sequentially (by order of recall or arrival at the clinic).
  For Phase I, enrollment was stopped once the goal of eight (8) subjects with xerostomia and eight (8) subjects without xerostomia has been reached.
  For Phase II, 16 subjects with xerostomia that were evaluated or treated at the clinic were enrolled sequentially (by order of recall or arrival at the clinic).
Pre-assignment Details: Period 1 was devoted to Phase I that included 8 subjects with and 8 without xerostomia.
  Period 2 was devoted to Phase II that included 16 subjects with xerostomia. Eight of those participated previously in Phase II.
Groups:
- Subjects With Xerostomia: Subjects complaining of xerostomia
- Subjects Without Xerostomia: Subjects not complaining of xerostomia
Period: Selection of the SaliPen Device
Arm/Group | Subjects With Xerostomia | Subjects Without Xerostomia
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Use of the SaliPen Device
Arm/Group | Subjects With Xerostomia | Subjects Without Xerostomia
Started (Participants of Arm I were the 8 subjects with xerostomia of Phase 1 and other 8 additional subjects with xerostomia. Arm II was not part of Phase II. Thus, none of the subjects without xerostomia of Phase I participated in Phase II) | 16 (Participants were the 8 subjects with xerostomia of Phase 1 and other 8 additional subjects with xerostomia) | 0 (None of the subjects without xerostomia of Phase I participated in Phase II)
Completed | 16 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In Phase I: Eight (8) 'All Comers' to an oral health clinic with no xerostomia and eight (8) patients with xerostomia.
  In Phase II: Sixteen (16) xerostomia patients (eight (8) of them participated in Phase I).
Groups:
- Selection and/or Use of the SaliPen Device by Subjects With or Without Xerostomia: Phase I Subjects with and without xerostomia were requested to read the label text on the outside of the study product package (external labeling) and determine whether the study product addresses their needs, without a provider direction or assistance.
  Phase II The study product was dispensed only to subjects with xerostomia. They were requested to use it with no training, except for their understanding of the User Manual (internal labeling). Those subjects used the study product in a supervised clinical setting.
Arm/Group | Selection and/or Use of the SaliPen Device by Subjects With or Without Xerostomia
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — Population: The row populations differs from the overall number since 8 subjects participated in both phases. Thus, 24 subjects were recruited. Eight participated only in Phase I, 8 participated only in Phase II and 8 participated in both phases.
  Participants
    Phase I subjects without xerostomia: number analyzed (Participants) | 8
    Phase I subjects without xerostomia: <=18 years | 0
    Phase I subjects without xerostomia: Between 18 and 65 years | 7
    Phase I subjects without xerostomia: >=65 years | 1
    Phase I subjects with xerostomia: number analyzed (Participants) | 8
    Phase I subjects with xerostomia: <=18 years | 0
    Phase I subjects with xerostomia: Between 18 and 65 years | 5
    Phase I subjects with xerostomia: >=65 years | 3
    Phase II subjects without xerostomia: number analyzed (Participants) | 0
    Phase II subjects with xerostomia: number analyzed (Participants) | 16
    Phase II subjects with xerostomia: <=18 years | 0
    Phase II subjects with xerostomia: Between 18 and 65 years | 13
    Phase II subjects with xerostomia: >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] — Population: The row populations differs from the overall number since 8 subjects participated in both phases. Thus, 24 subjects were recruited. Eight participated only in Phase I, 8 participated only in Phase II and 8 participated in both phases.
  years
    Phase I subjects without xerostomia: number analyzed (Participants) | 8
    Phase I subjects without xerostomia | 47 [33 to 65]
    Phase I subjects with xerostomia: number analyzed (Participants) | 8
    Phase I subjects with xerostomia | 58 [32 to 76]
    Phase II subjects without xerostomia: number analyzed (Participants) | 0
    Phase II subjects with xerostomia: number analyzed (Participants) | 16
    Phase II subjects with xerostomia | 53 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The row populations differs from the overall number since 8 subjects participated in both phases. Thus, 24 subjects were recruited. Eight participated only in Phase I, 8 participated only in Phase II and 8 participated in both phases.
  Participants
    Phase I subjects without xerostomia: number analyzed (Participants) | 8
    Phase I subjects without xerostomia: Female | 4
    Phase I subjects without xerostomia: Male | 4
    Phase I subjects with xerostomia: number analyzed (Participants) | 8
    Phase I subjects with xerostomia: Female | 6
    Phase I subjects with xerostomia: Male | 2
    Phase II subjects without xerostomia: number analyzed (Participants) | 0
    Phase II subjects with xerostomia: number analyzed (Participants) | 16
    Phase II subjects with xerostomia: Female | 14
    Phase II subjects with xerostomia: Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The row populations differs from the overall number since 8 subjects participated in both phases. Thus, 24 subjects were recruited. Eight participated only in Phase I, 8 participated only in Phase II and 8 participated in both phases.
  Participants
    Phase I subjects without xerostomia: number analyzed (Participants) | 8
    Phase I subjects without xerostomia: American Indian or Alaska Native | 0
    Phase I subjects without xerostomia: Asian | 4
    Phase I subjects without xerostomia: Native Hawaiian or Other Pacific Islander | 0
    Phase I subjects without xerostomia: Black or African American | 1
    Phase I subjects without xerostomia: White | 3
    Phase I subjects without xerostomia: More than one race | 0
    Phase I subjects without xerostomia: Unknown or Not Reported | 0
    Phase I subjects with xerostomia: number analyzed (Participants) | 8
    Phase I subjects with xerostomia: American Indian or Alaska Native | 0
    Phase I subjects with xerostomia: Asian | 0
    Phase I subjects with xerostomia: Native Hawaiian or Other Pacific Islander | 0
    Phase I subjects with xerostomia: Black or African American | 0
    Phase I subjects with xerostomia: White | 7
    Phase I subjects with xerostomia: More than one race | 1
    Phase I subjects with xerostomia: Unknown or Not Reported | 0
    Phase II subjects without xerostomia: number analyzed (Participants) | 0
    Phase II subjects with xerostomia: number analyzed (Participants) | 16
    Phase II subjects with xerostomia: American Indian or Alaska Native | 0
    Phase II subjects with xerostomia: Asian | 0
    Phase II subjects with xerostomia: Native Hawaiian or Other Pacific Islander | 0
    Phase II subjects with xerostomia: Black or African American | 0
    Phase II subjects with xerostomia: White | 14
    Phase II subjects with xerostomia: More than one race | 2
    Phase II subjects with xerostomia: Unknown or Not Reported | 0
Xerostomia status based on self-report (suffering or not from xerostomia) [Count of Participants; unit: Participants] — Xerostomia status was determined through self-report. Subjects attending the clinic were asked whether they suffer or not from xerostomia. According to their answer, they were allocated to each group: subjects with xerostomia or subjects without xerostomia. Population: Overall participant number was 24. 8 (with no xerostomia) participated only in Phase I . 8 (with xerostomia) participated only in Phase II. 8 (with xerostomia) participated in both, Phase I and Phase II.
  Participants
    Phase I subjects without xerostomia: number analyzed (Participants) | 8
    Phase I subjects without xerostomia | 8
    Phase I subjects with xerostomia: number analyzed (Participants) | 8
    Phase I subjects with xerostomia | 8
    Phase II subjects without xerostomia: number analyzed (Participants) | 0
    Phase II subjects with xerostomia: number analyzed (Participants) | 16
    Phase II subjects with xerostomia | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Appropriately Will Self-select the Study Product for Use Under Simulated OTC Conditions [Phase I]
Description: Following the standard norms for the Rx-to-OTC switch process, this outcome is a validation of potential consumers' ability to self-diagnose the condition and to decide that treatment with the product is appropriate for them.
Time Frame: One hour
Population: Eight subjects with xerostomia and 8 subjects without xerostomia
Measure: Number; unit: percentage
Groups:
- Experimental: Use of SaliPen Medical Device: Allocation to this group according to self-decision.
Arm/Group | Experimental: Use of SaliPen Medical Device
Number analyzed (Participants) | 16
percentage
  Percentage of correct answers to the question on eligibility to use the SaliPen device | 100
  Percentage of patients providing correct answers | 100

2. Primary Outcome: Percentage of Participants Who Correctly Will Use the Study Product When Dispensed Under Simulated OTC Conditions [Phase II].
Description: Correct use means that the participants will demonstrate the use of the study product according to the guidelines outlined in the User Manual.
  Following the standard norms for the therapy of Rx-to-OTC switch process, this outcome is a validation of potential consumers' ability to self-treat with the product according to the product's supplied IFU.
Time Frame: 1.5 hour
Population: All patients suffered from xerostomia
Measure: Number; unit: percentage
Arm/Group | Experimental: Use of SaliPen Medical Device
Number analyzed (Participants) | 16
percentage
  Percentage of correct performances | 100
  Percentage of subjects performing correctly | 100

ADVERSE EVENTS:
Time Frame: 1 month
Description: The examiners observed the occurrence of any adverse events.
Groups:
- Phase I: Selection of the SaliPen Device by Subjects With or Without Xerostomia: Subjects with and without xerostomia were requested to read the label text on the outside of the study product package (external labeling) and determine whether the study product addresses their needs, without a provider direction or assistance.
- Phase II: Use of the SaliPen Device by Subjects With Xerostomia: The study product was dispensed only to subjects with xerostomia. They were requested to use it with no training, except for their understanding of the User Manual (internal labeling). Those subjects used the study product in a supervised clinical setting.
Arm/Group | Phase I: Selection of the SaliPen Device by Subjects With or Without Xerostomia | Phase II: Use of the SaliPen Device by Subjects With Xerostomia
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT05058430/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT05058430/ICF_001.pdf